CLINICAL TRIAL: NCT01051804
Title: Evaluation of the Repeated Usage of Systane Ultra Eyedrop
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SMA-09-33
Record Dates: First submitted 2010-01-18; First posted 2010-01-20 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-01

CONDITIONS: Dry Eye
Keywords: Dry eye; Visual Performance
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Systane Ultra (Experimental): Systane Ultra Lubricant Eye Drops
  Interventions: Other: Systane Ultra
- Optive (Active Comparator): Optive Lubricant Eye Drops
  Interventions: Other: Optive lubricant Eye Drops

INTERVENTIONS:
Other: Systane Ultra — Systane Ultra 1 to 2 drops per eye at least 4 times daily for 4 weeks
  Arms: Systane Ultra
Other: Optive lubricant Eye Drops — Optive Lubricant Eye Drops 1 to 2 drops per eye at least 4 times daily for 4 weeks
  Arms: Optive

SUMMARY:
Comparison of two contact lens solutions.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or more.
* Non contact lens wearer.
* Symptomatology as defined below for the Ocular Surface Disease Index (OSDI) questionnaire:

  * Score ≥13 for OSDI Questionnaire total score; AND
  * Scores of at least 2 for 2 out of the 6 vision related questions of the OSDI questionnaire
* Best visual acuity of 6/9 or better in each eye.
* Willingness to adhere to the instructions set in the clinical protocol.
* Signature of the subject informed consent form.

Exclusion Criteria:

* Use of systemic medication which might produce dry eye side effects.
* Systemic disease which might produce dry eye side effects.
* Active ocular infection.
* Use of ocular medication.
* Significant ocular anomaly.
* Previous ocular surgery
* Previous use of Restasis
* Any medical condition that might be prejudicial to the study.
* The subject, based on their knowledge, must NOT be pregnant or lactating at the time of enrolment.
* The subject, based on his/her knowledge, must NOT have an infectious disease (e.g. hepatitis, tuberculosis) or an immunosuppressive disease (e.g. Human Immunodeficiency Virus).
* The subject, based on their knowledge, must NOT have diabetes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2009-11; Primary Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Improvement in objective vision | 4 weeks

SECONDARY OUTCOMES:
Measurement of tear film evaporation | 4 weeks